CLINICAL TRIAL: NCT07260877
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study With an Open-Label Extension Evaluating the Efficacy and Safety of VENT-03 in Adult Participants With Active Cutaneous Lupus Erythematosus With or Without Systemic Lupus Erythematosus
Acronym: AERIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ventus Therapeutics U.S., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VENT-03-201; 2024-520098-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-10; First posted 2025-12-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Lupus Erythematosus (CLE); Systemic Lupus Erythematosus; SLE; SLE (Systemic Lupus); CLE
Keywords: CLE, SLE, lupus, cutaneous lupus erythematosus, systemic lupus erythematosus, VENT-03; cGAS
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VENT-03 (Experimental): VENT-03
  Interventions: Drug: VENT-03
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VENT-03 — VENT-03 is a tablet
  Arms: VENT-03
Drug: Placebo — Placebo is a tablet
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if VENT-03 works to treat patients with cutaneous lupus erythematosus (CLE) who may or may not have systemic lupus erythematosus (SLE). Another goal is to learn about the safety of VENT-03 and how it is processed by the body. The main questions it aims to answer are:

* Does VENT-03 affect the activity and severity of CLE?
* What side effects do participants have when taking VENT-03?

Researchers will compare VENT-03 to a placebo (a look-alike substance that contains no drug) to see if VENT-03 works to treat patients with CLE.

Participants will:

* Take VENT-03 or a placebo e for 4 weeks, then all participants will switch to VENT-03 for another 8 weeks;
* Visit the clinic once a month for checkups and tests.

ELIGIBILITY:
Key Inclusion Criteria:

* Cutaneous lupus:

  * CLASI-A score ≥8;
  * At least 1 active discoid lupus erythematosus (DLE) lesion, OR at least 1 active subacute CLE lesion
* If participant has previous SLE diagnosis:

  * Positive antinuclear antibody test at Screening by immunofluorescent assay at the central laboratory with titer ≥ 1:80;
  * Meets the American College of Rheumatology/ European Alliance of Associations for Rheumatology 2019 criteria for SLE; and
  * Currently receiving at least one of the specified SLE medication treatments, at stable doses.

Key Exclusion Criteria:

* Meet protocol-specified infection or lab criteria; any other laboratory test results that, in the investigator's opinion, might place participant at unacceptable risk for participating in this study;
* Moderate or severe liver impairment as classified by the Child-Pugh criteria (categories B and C);
* Has drug-induced lupus, rather than 'idiopathic' lupus;
* History of, or current, inflammatory joint or skin disease other than SLE and cutaneous lupus;
* Diagnosis of select potentially confounding autoimmune disorders
* Active severe or unstable neuropsychiatric SLE;
* Hospitalization for a severe lupus flare in the past 3 months, or active severe SLE-driven disease, including lupus nephritis, for which in the opinion of the PI the protocol-specified SOC is insufficient;
* History of or current diagnosis of anti-phospholipid syndrome;
* History of any non-lupus disease that has required treatment with oral or parenteral corticosteroids for more than a total of 2 weeks within the last 24 weeks prior to Day 1;
* Meets protocol specified medical history of infectious diseases and infections and/or opportunistic infection requiring hospitalization or parenteral antimicrobial treatment within specified timeframes;
* Cancer screening results suspicious of malignancy or history of cancer within time specified with exceptions for curative therapy for squamous or basil cell carcinoma and cervical cancer in situ; and
* Meets protocol specified exclusions related to concomitant medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of VENT-03 on the interferon gene signature in the skin | Baseline to End of Double-Blind Treatment (up to Day 28)
  Percent change from baseline in interferon gene signature in the skin at Day 28

SECONDARY OUTCOMES:
Evaluate the effect of VENT-03 on CLE disease severity | Baseline to End of Double-Blind Treatment (up to Day 28)
  Percent change from baseline in CLASI-A score at Day 28
Evaluate effect of VENT-03 on CLE disease severity | Baseline to End of Double-Blind Treatment (up to Day 28)
  Percentage of participants achieving CLASI-A 50 response (≥ 50% improvement in CLASI A score compared with baseline) at Day 28
Change from Baseline in Myxovirus-Resistant Protein A (MXA) Immunostaining in Skin Biopsy | Baseline to End of Treatment (up to Day 84)
Number of participants with at least one Treatment Emergent Adverse Event (TEAE) and/or Serious Adverse Event (SAE) | Baseline to End of Treatment (up to Day 84)
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug. An SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of participants with Moderate or Severe Treatment Emergent Adverse Events (TEAEs) | Baseline to End of Treatment (up to Day 84)
Percentage of Participants with ≥ 1 Treatment Emergent Adverse Event (AE) leading to Treatment Discontinuation | Baseline to End of Treatment (up to Day 84)
Cmax: Maximum Observed Plasma Concentration for VENT-03 | Day 1 pre-dose and at multiple time points (up to 6 hours) post-dose; Day 28 pre-dose and post-dose; Day 56 and Day 84 pre-dose
AUClast: Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration for VENT-03 | Day 1 pre-dose and at multiple time points (up to 6 hours) post-dose; Day 28 pre-dose and post-dose; Day 56 and Day 84 pre-dose

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Investigative Site, Beverly Hills, California
  - Investigative Site, Clearwater, Florida
  - Investigative Site, DeBary, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Saint Joseph, Missouri
  - Investigative Site, Fairport, New York
  - Investigative Site, Memphis, Tennessee
  - Investigative Site, Allen, Texas
  - Investigative Site, Arlington, Texas
  - Investigative Site, Colleyville, Texas

IPD SHARING:
Plan to Share IPD: Undecided
As this study will enroll patients from the EU, the sponsor needs to consider that an IPD plan is compliant with GDPR. The sponsor needs to analyze and determine whether an IPD Plan can comply with GDPR based on plans and processes in place for the study in order to ensure legality and ethical data handling.